CLINICAL TRIAL: NCT00292552
Title: A Multicentre 3 Year Longitudinal Prospective Study to Identify Novel Endpoints and Compare These With Forced Expiratory Volume in 1 Second (FEV1) for Their Ability to Measure and Predict COPD Severity and Its Progression Over Time
Brief Title: Evaluation of COPD (Chronic Obstructive Pulmonary Disease) to Longitudinally Identify Predictive Surrogate Endpoints
Acronym: ECLIPSE
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: SCO104960
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD); longitudinal; eclipse
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, urine sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- COPD subjects: Subjects with GOLD stage II-IV COPD
  Interventions: Other: Novel endpoint determination
- Smoker controls: Subjects with smoking history but normal lung function
  Interventions: Other: Novel endpoint determination
- Non-smoker controls: Normal healthy non-smokers
  Interventions: Other: Novel endpoint determination

INTERVENTIONS:
Other: Novel endpoint determination — Novel endpoint determination

SUMMARY:
This is a 3 year longitudinal study to identify novel endpoints and compare these with standard measures such as forced expiratory volume in 1 second (FEV1) for their ability to measure and predict COPD (Chronic Obstructive Pulmonary Disease) severity and its progression over time. Control subjects (smokers and never smokers) will be recruited as comparators with the COPD subjects.

ELIGIBILITY:
Inclusion criteria:

* COPD Subjects
* A COPD subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Male or female subjects, aged 40-75 years inclusive
* A baseline (post-bronchodilator) FEV1 <80% of predicted normal and a baseline (post-bronchodilator) FEV1/FVC ratio 70%
* Current or ex-smokers with a smoking history of at least 10 pack-years (number of pack years = (number of cigarettes per day / 20) x number of years smoked e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years).
* A signed and dated written informed consent is obtained prior to participation
* Able to comply with the requirements of the protocol and be available for study visits over 3 years

Control Subjects - Current/Ex Smokers

* A control subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Male or female subjects, aged 40-75 years inclusive, who are free from significant disease as determined by history, physical examination and screening investigations
* Baseline (post-bronchodilator) FEV1 >85% of predicted normal. FEV1/FVC ratio >70%
* Current or ex-smokers with a smoking history of at least 10 pack-years (number of pack years = (number of cigarettes per day / 20) x number of years smoked e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years).
* A signed and dated written informed consent is obtained prior to participation.
* Able to comply with the requirements of the protocol and be available for study visits over 3 years

Control Subjects - Non-smokers

* A non-smoking control subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Male or female subjects, aged 40-75 years inclusive, who are free from significant disease as determined by history, physical examination and screening investigations
* Baseline (post-bronchodilator) FEV1 >85% of predicted normal. FEV1/FVC ratio >70%
* Non-smokers with a smoking history of < 1 pack-year (number of pack years = (number of cigarettes per day / 20) x number of years smoked).
* A signed and dated written informed consent is obtained prior to participation.
* Able to comply with the requirements of the protocol and be available for study visits over 3 years

Exclusion Criteria:

COPD Subjects

* A COPD subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Known respiratory disorders, or disorders identified at screening/visit 1 (including identification on the first CT scan), other than COPD (e.g.: lung cancer, sarcoidosis, tuberculosis, lung fibrosis, cystic fibrosis)
* Known history of significant inflammatory disease, other than COPD (e.g. rheumatoid arthritis and Lupus)
* Known to be severely alpha-1-antitrypsin deficient (PI SZ or ZZ)
* Having undergone lung surgery (e.g. lung reduction, lung transplant)
* Have cancer or have had cancer in the 5 years prior to study entry
* Serious, uncontrolled disease (including serious psychological disorders) likely to interfere with the study or impact on subject safety
* Is enrolled in a long term blinded drug study (subjects in open label studies may be considered and subjects in short blinded studies (approx less than 12 weeks may be considered following consultation with sponsor) or a study where there is significant radiation exposure (e.g.: CT scans)
* Have, in the opinion of the investigator, evidence of alcohol, drug or solvent abuse
* Have received a blood transfusion in the 4 weeks prior to study start
* Has experienced a moderate or severe exacerbation (requiring oral corticosteroid, antibiotics or hospitalisation) within the last 4 weeks. All courses of oral corticosteroids and antibiotics must be completed at least 2 weeks before study start
* Is on long term oral corticosteroids (long term is considered use for more than 3 consecutive months)
* Unable to walk
* Subject is a participating investigator, sub-investigator, study co-ordinator, or employee of a participating investigator, or is an immediate family member of the aforementioned.

Control Subjects

* A control subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Known respiratory disorders, or disorders identified at screening/visit 1 including identification on the first CT scan (e.g.: COPD, asthma, lung cancer, sarcoidosis, tuberculosis, lung fibrosis)
* Known history of significant inflammatory disease (eg rheumatoid arthritis and Lupus)
* Known to be severely alpha-1-antitrypsin deficient (PI SZ or ZZ)
* Having undergone lung surgery (e.g. lung reduction, lung transplant)
* Have cancer or have had cancer in the 5 years prior to study entry
* Serious, uncontrolled disease (including serious psychological disorders) likely to interfere with the study
* Is enrolled in a long term blinded drug study (subjects in open label studies may be considered and subjects in short blinded studies (approx less than 12 weeks may be considered following consultation with sponsor) or a study where there is significant radiation exposure (e.g.: CT scans)
* Have, in the opinion of the investigator, evidence of alcohol, drug or solvent abuse.
* Have received a blood transfusion in the 4 weeks prior to study start
* Is on long term oral corticosteroids (long term is considered use for more than 3 consecutive months)
* Subject is a participating investigator, sub-investigator, study co-ordinator, or employee of a participating investigator, or is an immediate family member of the aforementioned.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD subjects and smoking and non-smoking controls
Sampling Method: Probability Sample
Enrollment: 2747 (Actual)
Dates: Start 2005-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Identifying new patient subtypes and endpoints for COPD | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (18):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Richmond, Virginia
- Bulgaria (2):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Sofia
- Canada (6):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- GSK Investigational Site, Prague, Czechia
- GSK Investigational Site, Hvidovre, Denmark
- GSK Investigational Site, Horn, Netherlands
- GSK Investigational Site, Wellington, New Zealand
- GSK Investigational Site, Bergen, Norway
- GSK Investigational Site, Golnik, Slovenia
- GSK Investigational Site, Palma de Mallorca, Spain
- Ukraine (2):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kiev
- United Kingdom (5):
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

REFERENCES:
- [Derived] Zhang C, Konigsberg IR, He Y, Zhang J, Chikowore T, Feldman WB, Hu X, Ding Y, Pasaniuc B, Chang D, Chen Q, Lasky-Su JA, Hecker J, Tobin MD, Chen J, Kalra S, Pratte KA, Im HK, Wan ES, Manichaikul A, Silverman EK, Bowler RP, Lange LA, Ortega VE, Martin AR, Cho MH, Moll MR. Multi-Trait Polygenic Scores for COPD and COPD Exacerbations Implicate Druggable Proteins. medRxiv [Preprint]. 2025 Aug 26:2025.08.22.25334001. doi: 10.1101/2025.08.22.25334001. PMID 40909810
- [Derived] Suryadevara R, Gregory A, Lu R, Xu Z, Masoomi A, Lutz SM, Berman S, Yun JH, Saferali A, Ryu MH, Moll M, Sin DD, Hersh CP, Silverman EK, Dy J, Pratte KA, Bowler RP, Castaldi PJ, Boueiz A; COPDGene investigators. Blood-based Transcriptomic and Proteomic Biomarkers of Emphysema. Am J Respir Crit Care Med. 2024 Feb 1;209(3):273-287. doi: 10.1164/rccm.202301-0067OC. PMID 37917913
- [Derived] Govoni M, Bassi M, Santoro D, Donegan S, Singh D. Serum IL-8 as a Determinant of Response to Phosphodiesterase-4 Inhibition in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2023 Sep 1;208(5):559-569. doi: 10.1164/rccm.202301-0071OC. PMID 37192443
- [Derived] Hayden LP, Hobbs BD, Busch R, Cho MH, Liu M, Lopes-Ramos CM, Lomas DA, Bakke P, Gulsvik A, Silverman EK, Crapo JD, Beaty TH, Laird NM, Lange C, DeMeo DL. X chromosome associations with chronic obstructive pulmonary disease and related phenotypes: an X chromosome-wide association study. Respir Res. 2023 Feb 1;24(1):38. doi: 10.1186/s12931-023-02337-1. PMID 36726148
- [Derived] Mathur R, Fang F, Gaddis N, Hancock DB, Cho MH, Hokanson JE, Bierut LJ, Lutz SM, Young K, Smith AV; NHLBI Trans-Omics for Precision Medicine (TOPMed) Consortium; Silverman EK, Page GP, Johnson EO. GAWMerge expands GWAS sample size and diversity by combining array-based genotyping and whole-genome sequencing. Commun Biol. 2022 Aug 11;5(1):806. doi: 10.1038/s42003-022-03738-6. PMID 35953715
- [Derived] Driessen JHM, van Dort MJ, Romme EAPM, Wouters EFM, Smeenk FWJM, van Rietbergen B, van den Bergh JPW, Geusens P. Associations between bone attenuation and prevalent vertebral fractures on chest CT scans differ with vertebral fracture locations. Osteoporos Int. 2021 Sep;32(9):1869-1877. doi: 10.1007/s00198-020-05719-z. Epub 2021 Feb 16. PMID 33594489
- [Derived] Ash SY, San Jose Estepar R, Fain SB, Tal-Singer R, Stockley RA, Nordenmark LH, Rennard S, Han MK, Merrill D, Humphries SM, Diaz AA, Mason SE, Rahaghi FN, Pistenmaa CL, Sciurba FC, Vegas-Sanchez-Ferrero G, Lynch DA, Washko GR; COPDGene Investigators and the COPD Biomarker Qualification Consortium. Relationship between Emphysema Progression at CT and Mortality in Ever-Smokers: Results from the COPDGene and ECLIPSE Cohorts. Radiology. 2021 Apr;299(1):222-231. doi: 10.1148/radiol.2021203531. Epub 2021 Feb 16. PMID 33591891
- [Derived] Tang LYW, Coxson HO, Lam S, Leipsic J, Tam RC, Sin DD. Towards large-scale case-finding: training and validation of residual networks for detection of chronic obstructive pulmonary disease using low-dose CT. Lancet Digit Health. 2020 May;2(5):e259-e267. doi: 10.1016/S2589-7500(20)30064-9. Epub 2020 Apr 21. PMID 33328058
- [Derived] Celli B, Locantore N, Yates JC, Bakke P, Calverley PMA, Crim C, Coxson HO, Lomas DA, MacNee W, Miller BE, Mullerova H, Rennard SI, Silverman EK, Wouters E, Tal-Singer R, Agusti A, Vestbo J; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Markers of disease activity in COPD: an 8-year mortality study in the ECLIPSE cohort. Eur Respir J. 2021 Mar 25;57(3):2001339. doi: 10.1183/13993003.01339-2020. Print 2021 Mar. PMID 33303557
- [Derived] Moll M, Lutz SM, Ghosh AJ, Sakornsakolpat P, Hersh CP, Beaty TH, Dudbridge F, Tobin MD, Mittleman MA, Silverman EK, Hobbs BD, Cho MH. Relative contributions of family history and a polygenic risk score on COPD and related outcomes: COPDGene and ECLIPSE studies. BMJ Open Respir Res. 2020 Nov;7(1):e000755. doi: 10.1136/bmjresp-2020-000755. PMID 33239407
- [Derived] Langholm LL, Ronnow SR, Sand JMB, Leeming DJ, Tal-Singer R, Miller BE, Vestbo J, Karsdal MA, Manon-Jensen T. Increased von Willebrand Factor Processing in COPD, Reflecting Lung Epithelium Damage, Is Associated with Emphysema, Exacerbations and Elevated Mortality Risk. Int J Chron Obstruct Pulmon Dis. 2020 Mar 9;15:543-552. doi: 10.2147/COPD.S235673. eCollection 2020. PMID 32210548
- [Derived] Kim W, Cho MH, Sakornsakolpat P, Lynch DA, Coxson HO, Tal-Singer R, Silverman EK, Beaty TH. DSP variants may be associated with longitudinal change in quantitative emphysema. Respir Res. 2019 Jul 19;20(1):160. doi: 10.1186/s12931-019-1097-8. PMID 31324189
- [Derived] Ronnow SR, Sand JMB, Langholm LL, Manon-Jensen T, Karsdal MA, Tal-Singer R, Miller BE, Vestbo J, Leeming DJ. Type IV collagen turnover is predictive of mortality in COPD: a comparison to fibrinogen in a prospective analysis of the ECLIPSE cohort. Respir Res. 2019 Apr 1;20(1):63. doi: 10.1186/s12931-019-1026-x. PMID 30935391
- [Derived] Sakornsakolpat P, McCormack M, Bakke P, Gulsvik A, Make BJ, Crapo JD, Cho MH, Silverman EK. Genome-Wide Association Analysis of Single-Breath DlCO. Am J Respir Cell Mol Biol. 2019 May;60(5):523-531. doi: 10.1165/rcmb.2018-0384OC. PMID 30694715
- [Derived] Miller ER, Putman RK, Diaz AA, Xu H, San Jose Estepar R, Araki T, Nishino M, Poli de Frias S, Hida T, Ross J, Coxson H, Dupuis J, O'Connor GT, Silverman EK, Rosas IO, Hatabu H, Washko G, Hunninghake GM. Increased Airway Wall Thickness in Interstitial Lung Abnormalities and Idiopathic Pulmonary Fibrosis. Ann Am Thorac Soc. 2019 Apr;16(4):447-454. doi: 10.1513/AnnalsATS.201806-424OC. PMID 30543456
- [Derived] Naya IP, Tombs L, Muellerova H, Compton C, Jones PW. Long-term outcomes following first short-term clinically important deterioration in COPD. Respir Res. 2018 Nov 20;19(1):222. doi: 10.1186/s12931-018-0928-3. PMID 30453972
- [Derived] Boueiz A, Pham B, Chase R, Lamb A, Lee S, Naing ZZC, Cho MH, Parker MM, Sakornsakolpat P, Hersh CP, Crapo JD, Stergachis AB, Tal-Singer R, DeMeo DL, Silverman EK, Zhou X, Castaldi PJ; COPDGene investigators, by Core Units:, ECLIPSE Investigators:, GenKOLS Investigators:. Integrative Genomics Analysis Identifies ACVR1B as a Candidate Causal Gene of Emphysema Distribution. Am J Respir Cell Mol Biol. 2019 Apr;60(4):388-398. doi: 10.1165/rcmb.2018-0110OC. PMID 30335480
- [Derived] Sakornsakolpat P, Morrow JD, Castaldi PJ, Hersh CP, Bosse Y, Silverman EK, Manichaikul A, Cho MH. Integrative genomics identifies new genes associated with severe COPD and emphysema. Respir Res. 2018 Mar 22;19(1):46. doi: 10.1186/s12931-018-0744-9. PMID 29566699
- [Derived] Celli BR, Locantore N, Tal-Singer R, Riley J, Miller B, Vestbo J, Yates JC, Silverman EK, Owen CA, Divo M, Pinto-Plata V, Wouters EFM, Faner R, Agusti A; ECLIPSE Study Investigators. Emphysema and extrapulmonary tissue loss in COPD: a multi-organ loss of tissue phenotype. Eur Respir J. 2018 Feb 7;51(2):1702146. doi: 10.1183/13993003.02146-2017. Print 2018 Feb. PMID 29437944
- [Derived] Morrow JD, Cho MH, Platig J, Zhou X, DeMeo DL, Qiu W, Celli B, Marchetti N, Criner GJ, Bueno R, Washko GR, Glass K, Quackenbush J, Silverman EK, Hersh CP. Ensemble genomic analysis in human lung tissue identifies novel genes for chronic obstructive pulmonary disease. Hum Genomics. 2018 Jan 15;12(1):1. doi: 10.1186/s40246-018-0132-z. PMID 29335020
- [Derived] Obeidat M, Nie Y, Chen V, Shannon CP, Andiappan AK, Lee B, Rotzschke O, Castaldi PJ, Hersh CP, Fishbane N, Ng RT, McManus B, Miller BE, Rennard S, Pare PD, Sin DD. Network-based analysis reveals novel gene signatures in peripheral blood of patients with chronic obstructive pulmonary disease. Respir Res. 2017 Apr 24;18(1):72. doi: 10.1186/s12931-017-0558-1. PMID 28438154
- [Derived] Ishii T, Angata T, Wan ES, Cho MH, Motegi T, Gao C, Ohtsubo K, Kitazume S, Gemma A, ParE PD, Lomas DA, Silverman EK, Taniguchi N, Kida K. Influence of SIGLEC9 polymorphisms on COPD phenotypes including exacerbation frequency. Respirology. 2017 May;22(4):684-690. doi: 10.1111/resp.12952. Epub 2016 Nov 22. PMID 27878892
- [Derived] Sand JM, Leeming DJ, Byrjalsen I, Bihlet AR, Lange P, Tal-Singer R, Miller BE, Karsdal MA, Vestbo J. High levels of biomarkers of collagen remodeling are associated with increased mortality in COPD - results from the ECLIPSE study. Respir Res. 2016 Oct 4;17(1):125. doi: 10.1186/s12931-016-0440-6. PMID 27716343
- [Derived] Boueiz A, Lutz SM, Cho MH, Hersh CP, Bowler RP, Washko GR, Halper-Stromberg E, Bakke P, Gulsvik A, Laird NM, Beaty TH, Coxson HO, Crapo JD, Silverman EK, Castaldi PJ, DeMeo DL; COPDGene and ECLIPSE Investigators. Genome-Wide Association Study of the Genetic Determinants of Emphysema Distribution. Am J Respir Crit Care Med. 2017 Mar 15;195(6):757-771. doi: 10.1164/rccm.201605-0997OC. PMID 27669027
- [Derived] Huang JT, Bolton CE, Miller BE, Tal-Singer R, Rabinovich RA, Palmer CN, Thomson NC, MacNee W; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Age-dependent elastin degradation is enhanced in chronic obstructive pulmonary disease. Eur Respir J. 2016 Oct;48(4):1215-1218. doi: 10.1183/13993003.01125-2016. Epub 2016 Sep 1. No abstract available. PMID 27587547
- [Derived] Joppa P, Tkacova R, Franssen FM, Hanson C, Rennard SI, Silverman EK, McDonald ML, Calverley PM, Tal-Singer R, Spruit MA, Kenn K, Wouters EF, Rutten EP. Sarcopenic Obesity, Functional Outcomes, and Systemic Inflammation in Patients With Chronic Obstructive Pulmonary Disease. J Am Med Dir Assoc. 2016 Aug 1;17(8):712-8. doi: 10.1016/j.jamda.2016.03.020. Epub 2016 May 5. PMID 27161848
- [Derived] Obeidat M, Ding X, Fishbane N, Hollander Z, Ng RT, McManus B, Tebbutt SJ, Miller BE, Rennard S, Pare PD, Sin DD. The Effect of Different Case Definitions of Current Smoking on the Discovery of Smoking-Related Blood Gene Expression Signatures in Chronic Obstructive Pulmonary Disease. Nicotine Tob Res. 2016 Sep;18(9):1903-9. doi: 10.1093/ntr/ntw129. Epub 2016 May 6. PMID 27154971
- [Derived] Rabinovich RA, Miller BE, Wrobel K, Ranjit K, Williams MC, Drost E, Edwards LD, Lomas DA, Rennard SI, Agusti A, Tal-Singer R, Vestbo J, Wouters EF, John M, van Beek EJ, Murchison JT, Bolton CE, MacNee W, Huang JT; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Circulating desmosine levels do not predict emphysema progression but are associated with cardiovascular risk and mortality in COPD. Eur Respir J. 2016 May;47(5):1365-73. doi: 10.1183/13993003.01824-2015. Epub 2016 Mar 23. PMID 27009168
- [Derived] Wurst KE, Rheault TR, Edwards L, Tal-Singer R, Agusti A, Vestbo J. A comparison of COPD patients with and without ACOS in the ECLIPSE study. Eur Respir J. 2016 May;47(5):1559-62. doi: 10.1183/13993003.02045-2015. Epub 2016 Mar 17. No abstract available. PMID 26989103
- [Derived] Putman RK, Hatabu H, Araki T, Gudmundsson G, Gao W, Nishino M, Okajima Y, Dupuis J, Latourelle JC, Cho MH, El-Chemaly S, Coxson HO, Celli BR, Fernandez IE, Zazueta OE, Ross JC, Harmouche R, Estepar RS, Diaz AA, Sigurdsson S, Gudmundsson EF, Eiriksdottir G, Aspelund T, Budoff MJ, Kinney GL, Hokanson JE, Williams MC, Murchison JT, MacNee W, Hoffmann U, O'Donnell CJ, Launer LJ, Harrris TB, Gudnason V, Silverman EK, O'Connor GT, Washko GR, Rosas IO, Hunninghake GM; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators; COPDGene Investigators. Association Between Interstitial Lung Abnormalities and All-Cause Mortality. JAMA. 2016 Feb 16;315(7):672-81. doi: 10.1001/jama.2016.0518. PMID 26881370
- [Derived] Yohannes AM, Mullerova H, Hanania NA, Lavoie K, Tal-Singer R, Vestbo J, Rennard SI, Wouters EF. Long-term Course of Depression Trajectories in Patients With COPD: A 3-Year Follow-up Analysis of the Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints Cohort. Chest. 2016 Apr;149(4):916-26. doi: 10.1016/j.chest.2015.10.081. Epub 2016 Jan 5. PMID 26836938
- [Derived] Chang Y, Glass K, Liu YY, Silverman EK, Crapo JD, Tal-Singer R, Bowler R, Dy J, Cho M, Castaldi P. COPD subtypes identified by network-based clustering of blood gene expression. Genomics. 2016 Mar;107(2-3):51-58. doi: 10.1016/j.ygeno.2016.01.004. Epub 2016 Jan 8. PMID 26773458
- [Derived] Lutz SM, Cho MH, Young K, Hersh CP, Castaldi PJ, McDonald ML, Regan E, Mattheisen M, DeMeo DL, Parker M, Foreman M, Make BJ, Jensen RL, Casaburi R, Lomas DA, Bhatt SP, Bakke P, Gulsvik A, Crapo JD, Beaty TH, Laird NM, Lange C, Hokanson JE, Silverman EK; ECLIPSE Investigators; COPDGene Investigators. A genome-wide association study identifies risk loci for spirometric measures among smokers of European and African ancestry. BMC Genet. 2015 Dec 3;16:138. doi: 10.1186/s12863-015-0299-4. PMID 26634245
- [Derived] Exuzides A, Colby C, Briggs AH, Lomas DA, Rutten-van Molken MPMH, Tabberer M, Chambers M, Muellerova H, Locantore N, Risebrough NA, Ismaila AS, Gonzalez-McQuire S. Statistical Modeling of Disease Progression for Chronic Obstructive Pulmonary Disease Using Data from the ECLIPSE Study. Med Decis Making. 2017 May;37(4):453-468. doi: 10.1177/0272989X15610781. Epub 2015 Oct 8. PMID 26449490
- [Derived] Cho MH, Castaldi PJ, Hersh CP, Hobbs BD, Barr RG, Tal-Singer R, Bakke P, Gulsvik A, San Jose Estepar R, Van Beek EJ, Coxson HO, Lynch DA, Washko GR, Laird NM, Crapo JD, Beaty TH, Silverman EK; NETT Genetics, ECLIPSE, and COPDGene Investigators. A Genome-Wide Association Study of Emphysema and Airway Quantitative Imaging Phenotypes. Am J Respir Crit Care Med. 2015 Sep 1;192(5):559-69. doi: 10.1164/rccm.201501-0148OC. PMID 26030696
- [Derived] Wilke S, Jones PW, Mullerova H, Vestbo J, Tal-Singer R, Franssen FM, Agusti A, Bakke P, Calverley PM, Coxson HO, Crim C, Edwards LD, Lomas DA, MacNee W, Rennard SI, Yates JC, Wouters EF, Spruit MA. One-year change in health status and subsequent outcomes in COPD. Thorax. 2015 May;70(5):420-5. doi: 10.1136/thoraxjnl-2014-205697. Epub 2015 Mar 17. PMID 25782757
- [Derived] Rennard SI, Locantore N, Delafont B, Tal-Singer R, Silverman EK, Vestbo J, Miller BE, Bakke P, Celli B, Calverley PM, Coxson H, Crim C, Edwards LD, Lomas DA, MacNee W, Wouters EF, Yates JC, Coca I, Agusti A; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints. Identification of five chronic obstructive pulmonary disease subgroups with different prognoses in the ECLIPSE cohort using cluster analysis. Ann Am Thorac Soc. 2015 Mar;12(3):303-12. doi: 10.1513/AnnalsATS.201403-125OC. PMID 25642832
- [Derived] Mullerova H, Maselli DJ, Locantore N, Vestbo J, Hurst JR, Wedzicha JA, Bakke P, Agusti A, Anzueto A. Hospitalized exacerbations of COPD: risk factors and outcomes in the ECLIPSE cohort. Chest. 2015 Apr;147(4):999-1007. doi: 10.1378/chest.14-0655. PMID 25356881
- [Derived] Hersh CP, Make BJ, Lynch DA, Barr RG, Bowler RP, Calverley PM, Castaldi PJ, Cho MH, Coxson HO, DeMeo DL, Foreman MG, Han MK, Harshfield BJ, Hokanson JE, Lutz S, Ramsdell JW, Regan EA, Rennard SI, Schroeder JD, Sciurba FC, Steiner RM, Tal-Singer R, van Beek E Jr, Silverman EK, Crapo JD; COPDGene and ECLIPSE Investigators. Non-emphysematous chronic obstructive pulmonary disease is associated with diabetes mellitus. BMC Pulm Med. 2014 Oct 24;14:164. doi: 10.1186/1471-2466-14-164. PMID 25341556
- [Derived] Singh D, Kolsum U, Brightling CE, Locantore N, Agusti A, Tal-Singer R; ECLIPSE investigators. Eosinophilic inflammation in COPD: prevalence and clinical characteristics. Eur Respir J. 2014 Dec;44(6):1697-700. doi: 10.1183/09031936.00162414. Epub 2014 Oct 16. No abstract available. PMID 25323230
- [Derived] Lee JH, Cho MH, Hersh CP, McDonald ML, Crapo JD, Bakke PS, Gulsvik A, Comellas AP, Wendt CH, Lomas DA, Kim V, Silverman EK; COPDGene and ECLIPSE Investigators. Genetic susceptibility for chronic bronchitis in chronic obstructive pulmonary disease. Respir Res. 2014 Sep 21;15(1):113. doi: 10.1186/s12931-014-0113-2. PMID 25241909
- [Derived] Lee JH, McDonald ML, Cho MH, Wan ES, Castaldi PJ, Hunninghake GM, Marchetti N, Lynch DA, Crapo JD, Lomas DA, Coxson HO, Bakke PS, Silverman EK, Hersh CP; COPDGene and ECLIPSE Investigators. DNAH5 is associated with total lung capacity in chronic obstructive pulmonary disease. Respir Res. 2014 Aug 20;15(1):97. doi: 10.1186/s12931-014-0097-y. PMID 25134640
- [Derived] Menche J, Sharma A, Cho MH, Mayer RJ, Rennard SI, Celli B, Miller BE, Locantore N, Tal-Singer R, Ghosh S, Larminie C, Bradley G, Riley JH, Agusti A, Silverman EK, Barabasi AL. A diVIsive Shuffling Approach (VIStA) for gene expression analysis to identify subtypes in Chronic Obstructive Pulmonary Disease. BMC Syst Biol. 2014;8 Suppl 2(Suppl 2):S8. doi: 10.1186/1752-0509-8-S2-S8. Epub 2014 Mar 13. PMID 25032995
- [Derived] Wells JM, O'Reilly PJ, Szul T, Sullivan DI, Handley G, Garrett C, McNicholas CM, Roda MA, Miller BE, Tal-Singer R, Gaggar A, Rennard SI, Jackson PL, Blalock JE. An aberrant leukotriene A4 hydrolase-proline-glycine-proline pathway in the pathogenesis of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 Jul 1;190(1):51-61. doi: 10.1164/rccm.201401-0145OC. PMID 24874071
- [Derived] Vestbo J, Agusti A, Wouters EF, Bakke P, Calverley PM, Celli B, Coxson H, Crim C, Edwards LD, Locantore N, Lomas DA, MacNee W, Miller B, Rennard SI, Silverman EK, Yates JC, Tal-Singer R; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints Study Investigators. Should we view chronic obstructive pulmonary disease differently after ECLIPSE? A clinical perspective from the study team. Am J Respir Crit Care Med. 2014 May 1;189(9):1022-30. doi: 10.1164/rccm.201311-2006PP. PMID 24552242
- [Derived] Coxson HO, Dirksen A, Edwards LD, Yates JC, Agusti A, Bakke P, Calverley PM, Celli B, Crim C, Duvoix A, Fauerbach PN, Lomas DA, Macnee W, Mayer RJ, Miller BE, Muller NL, Rennard SI, Silverman EK, Tal-Singer R, Wouters EF, Vestbo J; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. The presence and progression of emphysema in COPD as determined by CT scanning and biomarker expression: a prospective analysis from the ECLIPSE study. Lancet Respir Med. 2013 Apr;1(2):129-36. doi: 10.1016/S2213-2600(13)70006-7. Epub 2013 Feb 1. PMID 24429093
- [Derived] Cheng DT, Kim DK, Cockayne DA, Belousov A, Bitter H, Cho MH, Duvoix A, Edwards LD, Lomas DA, Miller BE, Reynaert N, Tal-Singer R, Wouters EF, Agusti A, Fabbri LM, Rames A, Visvanathan S, Rennard SI, Jones P, Parmar H, MacNee W, Wolff G, Silverman EK, Mayer RJ, Pillai SG; TESRA and ECLIPSE Investigators. Systemic soluble receptor for advanced glycation endproducts is a biomarker of emphysema and associated with AGER genetic variants in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2013 Oct 15;188(8):948-57. doi: 10.1164/rccm.201302-0247OC. PMID 23947473
- [Derived] Ubhi BK, Davenport PW, Welch M, Riley J, Griffin JL, Connor SC. Analysis of chloroformate-derivatised amino acids, dipeptides and polyamines by LC-MS/MS. J Chromatogr B Analyt Technol Biomed Life Sci. 2013 Sep 1;934:79-88. doi: 10.1016/j.jchromb.2013.06.026. Epub 2013 Jun 29. PMID 23911539
- [Derived] Donaldson GC, Mullerova H, Locantore N, Hurst JR, Calverley PM, Vestbo J, Anzueto A, Wedzicha JA. Factors associated with change in exacerbation frequency in COPD. Respir Res. 2013 Jul 30;14(1):79. doi: 10.1186/1465-9921-14-79. PMID 23899210
- [Derived] Berg I, Hanson C, Sayles H, Romberger D, Nelson A, Meza J, Miller B, Wouters EF, Macnee W, Rutten EP, Romme EA, Vestbo J, Edwards L, Rennard S. Vitamin D, vitamin D binding protein, lung function and structure in COPD. Respir Med. 2013 Oct;107(10):1578-88. doi: 10.1016/j.rmed.2013.05.010. Epub 2013 Jul 1. PMID 23809536
- [Derived] Sumner H, Woodcock A, Kolsum U, Dockry R, Lazaar AL, Singh D, Vestbo J, Smith JA. Predictors of objective cough frequency in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2013 May 1;187(9):943-9. doi: 10.1164/rccm.201211-2000OC. PMID 23471467
- [Derived] Zhou X, Qiu W, Sathirapongsasuti JF, Cho MH, Mancini JD, Lao T, Thibault DM, Litonjua AA, Bakke PS, Gulsvik A, Lomas DA, Beaty TH, Hersh CP, Anderson C, Geigenmuller U, Raby BA, Rennard SI, Perrella MA, Choi AM, Quackenbush J, Silverman EK. Gene expression analysis uncovers novel hedgehog interacting protein (HHIP) effects in human bronchial epithelial cells. Genomics. 2013 May;101(5):263-72. doi: 10.1016/j.ygeno.2013.02.010. Epub 2013 Mar 1. PMID 23459001
- [Derived] Kim DK, Cho MH, Hersh CP, Lomas DA, Miller BE, Kong X, Bakke P, Gulsvik A, Agusti A, Wouters E, Celli B, Coxson H, Vestbo J, MacNee W, Yates JC, Rennard S, Litonjua A, Qiu W, Beaty TH, Crapo JD, Riley JH, Tal-Singer R, Silverman EK; ECLIPSE, ICGN, and COPDGene Investigators. Genome-wide association analysis of blood biomarkers in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2012 Dec 15;186(12):1238-47. doi: 10.1164/rccm.201206-1013OC. Epub 2012 Nov 9. PMID 23144326
- [Derived] Ubhi BK, Cheng KK, Dong J, Janowitz T, Jodrell D, Tal-Singer R, MacNee W, Lomas DA, Riley JH, Griffin JL, Connor SC. Targeted metabolomics identifies perturbations in amino acid metabolism that sub-classify patients with COPD. Mol Biosyst. 2012 Oct 30;8(12):3125-33. doi: 10.1039/c2mb25194a. PMID 23051772
- [Derived] Wells JM, Washko GR, Han MK, Abbas N, Nath H, Mamary AJ, Regan E, Bailey WC, Martinez FJ, Westfall E, Beaty TH, Curran-Everett D, Curtis JL, Hokanson JE, Lynch DA, Make BJ, Crapo JD, Silverman EK, Bowler RP, Dransfield MT; COPDGene Investigators; ECLIPSE Study Investigators. Pulmonary arterial enlargement and acute exacerbations of COPD. N Engl J Med. 2012 Sep 6;367(10):913-21. doi: 10.1056/NEJMoa1203830. Epub 2012 Sep 3. PMID 22938715
- [Derived] Al-shair K, Muellerova H, Yorke J, Rennard SI, Wouters EF, Hanania NA, Sharafkhaneh A, Vestbo J; ECLIPSE investigators. Examining fatigue in COPD: development, validity and reliability of a modified version of FACIT-F scale. Health Qual Life Outcomes. 2012 Aug 23;10:100. doi: 10.1186/1477-7525-10-100. PMID 22913289
- [Derived] Wilk JB, Shrine NR, Loehr LR, Zhao JH, Manichaikul A, Lopez LM, Smith AV, Heckbert SR, Smolonska J, Tang W, Loth DW, Curjuric I, Hui J, Cho MH, Latourelle JC, Henry AP, Aldrich M, Bakke P, Beaty TH, Bentley AR, Borecki IB, Brusselle GG, Burkart KM, Chen TH, Couper D, Crapo JD, Davies G, Dupuis J, Franceschini N, Gulsvik A, Hancock DB, Harris TB, Hofman A, Imboden M, James AL, Khaw KT, Lahousse L, Launer LJ, Litonjua A, Liu Y, Lohman KK, Lomas DA, Lumley T, Marciante KD, McArdle WL, Meibohm B, Morrison AC, Musk AW, Myers RH, North KE, Postma DS, Psaty BM, Rich SS, Rivadeneira F, Rochat T, Rotter JI, Soler Artigas M, Starr JM, Uitterlinden AG, Wareham NJ, Wijmenga C, Zanen P, Province MA, Silverman EK, Deary IJ, Palmer LJ, Cassano PA, Gudnason V, Barr RG, Loos RJ, Strachan DP, London SJ, Boezen HM, Probst-Hensch N, Gharib SA, Hall IP, O'Connor GT, Tobin MD, Stricker BH. Genome-wide association studies identify CHRNA5/3 and HTR4 in the development of airflow obstruction. Am J Respir Crit Care Med. 2012 Oct 1;186(7):622-32. doi: 10.1164/rccm.201202-0366OC. Epub 2012 Jul 26. PMID 22837378
- [Derived] Albert P, Agusti A, Edwards L, Tal-Singer R, Yates J, Bakke P, Celli BR, Coxson HO, Crim C, Lomas DA, Macnee W, Miller B, Rennard S, Silverman EK, Vestbo J, Wouters E, Calverley P. Bronchodilator responsiveness as a phenotypic characteristic of established chronic obstructive pulmonary disease. Thorax. 2012 Aug;67(8):701-8. doi: 10.1136/thoraxjnl-2011-201458. Epub 2012 Jun 13. PMID 22696176
- [Derived] Agusti A, Edwards LD, Rennard SI, MacNee W, Tal-Singer R, Miller BE, Vestbo J, Lomas DA, Calverley PM, Wouters E, Crim C, Yates JC, Silverman EK, Coxson HO, Bakke P, Mayer RJ, Celli B; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Persistent systemic inflammation is associated with poor clinical outcomes in COPD: a novel phenotype. PLoS One. 2012;7(5):e37483. doi: 10.1371/journal.pone.0037483. Epub 2012 May 18. PMID 22624038
- [Derived] Celli BR, Locantore N, Yates J, Tal-Singer R, Miller BE, Bakke P, Calverley P, Coxson H, Crim C, Edwards LD, Lomas DA, Duvoix A, MacNee W, Rennard S, Silverman E, Vestbo J, Wouters E, Agusti A; ECLIPSE Investigators. Inflammatory biomarkers improve clinical prediction of mortality in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2012 May 15;185(10):1065-72. doi: 10.1164/rccm.201110-1792OC. Epub 2012 Mar 15. PMID 22427534
- [Derived] Waschki B, Spruit MA, Watz H, Albert PS, Shrikrishna D, Groenen M, Smith C, Man WD, Tal-Singer R, Edwards LD, Calverley PM, Magnussen H, Polkey MI, Wouters EF. Physical activity monitoring in COPD: compliance and associations with clinical characteristics in a multicenter study. Respir Med. 2012 Apr;106(4):522-30. doi: 10.1016/j.rmed.2011.10.022. Epub 2011 Nov 25. PMID 22118987
- [Derived] Cho MH, Castaldi PJ, Wan ES, Siedlinski M, Hersh CP, Demeo DL, Himes BE, Sylvia JS, Klanderman BJ, Ziniti JP, Lange C, Litonjua AA, Sparrow D, Regan EA, Make BJ, Hokanson JE, Murray T, Hetmanski JB, Pillai SG, Kong X, Anderson WH, Tal-Singer R, Lomas DA, Coxson HO, Edwards LD, MacNee W, Vestbo J, Yates JC, Agusti A, Calverley PM, Celli B, Crim C, Rennard S, Wouters E, Bakke P, Gulsvik A, Crapo JD, Beaty TH, Silverman EK; ICGN Investigators; ECLIPSE Investigators; COPDGene Investigators. A genome-wide association study of COPD identifies a susceptibility locus on chromosome 19q13. Hum Mol Genet. 2012 Feb 15;21(4):947-57. doi: 10.1093/hmg/ddr524. Epub 2011 Nov 11. PMID 22080838
- [Derived] Dickens JA, Miller BE, Edwards LD, Silverman EK, Lomas DA, Tal-Singer R; Evaluation of COPD Longitudinally to Identify Surrogate Endpoints (ECLIPSE) study investigators. COPD association and repeatability of blood biomarkers in the ECLIPSE cohort. Respir Res. 2011 Nov 4;12(1):146. doi: 10.1186/1465-9921-12-146. PMID 22054035
- [Derived] Vestbo J, Edwards LD, Scanlon PD, Yates JC, Agusti A, Bakke P, Calverley PM, Celli B, Coxson HO, Crim C, Lomas DA, MacNee W, Miller BE, Silverman EK, Tal-Singer R, Wouters E, Rennard SI; ECLIPSE Investigators. Changes in forced expiratory volume in 1 second over time in COPD. N Engl J Med. 2011 Sep 29;365(13):1184-92. doi: 10.1056/NEJMoa1105482. Epub 2011 Sep 26. PMID 21991892
- [Derived] Brehm JM, Hagiwara K, Tesfaigzi Y, Bruse S, Mariani TJ, Bhattacharya S, Boutaoui N, Ziniti JP, Soto-Quiros ME, Avila L, Cho MH, Himes B, Litonjua AA, Jacobson F, Bakke P, Gulsvik A, Anderson WH, Lomas DA, Forno E, Datta S, Silverman EK, Celedon JC. Identification of FGF7 as a novel susceptibility locus for chronic obstructive pulmonary disease. Thorax. 2011 Dec;66(12):1085-90. doi: 10.1136/thoraxjnl-2011-200017. Epub 2011 Sep 15. PMID 21921092
- [Derived] Spruit MA, Polkey MI, Celli B, Edwards LD, Watkins ML, Pinto-Plata V, Vestbo J, Calverley PM, Tal-Singer R, Agusti A, Coxson HO, Lomas DA, MacNee W, Rennard S, Silverman EK, Crim CC, Yates J, Wouters EF; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) study investigators. Predicting outcomes from 6-minute walk distance in chronic obstructive pulmonary disease. J Am Med Dir Assoc. 2012 Mar;13(3):291-7. doi: 10.1016/j.jamda.2011.06.009. Epub 2011 Jul 21. PMID 21778120
- [Derived] Siedlinski M, Cho MH, Bakke P, Gulsvik A, Lomas DA, Anderson W, Kong X, Rennard SI, Beaty TH, Hokanson JE, Crapo JD, Silverman EK; COPDGene Investigators; ECLIPSE Investigators. Genome-wide association study of smoking behaviours in patients with COPD. Thorax. 2011 Oct;66(10):894-902. doi: 10.1136/thoraxjnl-2011-200154. Epub 2011 Jun 16. PMID 21685187
- [Derived] Castaldi PJ, Cho MH, Litonjua AA, Bakke P, Gulsvik A, Lomas DA, Anderson W, Beaty TH, Hokanson JE, Crapo JD, Laird N, Silverman EK; COPDGene and Eclipse Investigators. The association of genome-wide significant spirometric loci with chronic obstructive pulmonary disease susceptibility. Am J Respir Cell Mol Biol. 2011 Dec;45(6):1147-53. doi: 10.1165/rcmb.2011-0055OC. Epub 2011 Jun 9. PMID 21659657
- [Derived] Crim C, Celli B, Edwards LD, Wouters E, Coxson HO, Tal-Singer R, Calverley PM; ECLIPSE investigators. Respiratory system impedance with impulse oscillometry in healthy and COPD subjects: ECLIPSE baseline results. Respir Med. 2011 Jul;105(7):1069-78. doi: 10.1016/j.rmed.2011.01.010. Epub 2011 Apr 11. PMID 21481577
- [Derived] Gietema HA, Muller NL, Fauerbach PV, Sharma S, Edwards LD, Camp PG, Coxson HO; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) investigators. Quantifying the extent of emphysema: factors associated with radiologists' estimations and quantitative indices of emphysema severity using the ECLIPSE cohort. Acad Radiol. 2011 Jun;18(6):661-71. doi: 10.1016/j.acra.2011.01.011. Epub 2011 Mar 9. PMID 21393027
- [Derived] Sin DD, Miller BE, Duvoix A, Man SF, Zhang X, Silverman EK, Connett JE, Anthonisen NA, Wise RA, Tashkin D, Celli BR, Edwards LD, Locantore N, Macnee W, Tal-Singer R, Lomas DA; ECLIPSE Investigators. Serum PARC/CCL-18 concentrations and health outcomes in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2011 May 1;183(9):1187-92. doi: 10.1164/rccm.201008-1220OC. Epub 2011 Jan 7. PMID 21216880
- [Derived] Hanania NA, Mullerova H, Locantore NW, Vestbo J, Watkins ML, Wouters EF, Rennard SI, Sharafkhaneh A; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) study investigators. Determinants of depression in the ECLIPSE chronic obstructive pulmonary disease cohort. Am J Respir Crit Care Med. 2011 Mar 1;183(5):604-11. doi: 10.1164/rccm.201003-0472OC. Epub 2010 Oct 1. PMID 20889909
- [Derived] Hurst JR, Vestbo J, Anzueto A, Locantore N, Mullerova H, Tal-Singer R, Miller B, Lomas DA, Agusti A, Macnee W, Calverley P, Rennard S, Wouters EF, Wedzicha JA; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Susceptibility to exacerbation in chronic obstructive pulmonary disease. N Engl J Med. 2010 Sep 16;363(12):1128-38. doi: 10.1056/NEJMoa0909883. PMID 20843247
- [Derived] Kong X, Cho MH, Anderson W, Coxson HO, Muller N, Washko G, Hoffman EA, Bakke P, Gulsvik A, Lomas DA, Silverman EK, Pillai SG; ECLIPSE Study NETT Investigators. Genome-wide association study identifies BICD1 as a susceptibility gene for emphysema. Am J Respir Crit Care Med. 2011 Jan 1;183(1):43-9. doi: 10.1164/rccm.201004-0541OC. Epub 2010 Aug 13. PMID 20709820
- [Derived] Singh D, Edwards L, Tal-Singer R, Rennard S. Sputum neutrophils as a biomarker in COPD: findings from the ECLIPSE study. Respir Res. 2010 Jun 15;11(1):77. doi: 10.1186/1465-9921-11-77. PMID 20550701
- [Derived] Cho MH, Boutaoui N, Klanderman BJ, Sylvia JS, Ziniti JP, Hersh CP, DeMeo DL, Hunninghake GM, Litonjua AA, Sparrow D, Lange C, Won S, Murphy JR, Beaty TH, Regan EA, Make BJ, Hokanson JE, Crapo JD, Kong X, Anderson WH, Tal-Singer R, Lomas DA, Bakke P, Gulsvik A, Pillai SG, Silverman EK. Variants in FAM13A are associated with chronic obstructive pulmonary disease. Nat Genet. 2010 Mar;42(3):200-2. doi: 10.1038/ng.535. Epub 2010 Feb 21. PMID 20173748
- [Derived] Lomas DA, Silverman EK, Edwards LD, Locantore NW, Miller BE, Horstman DH, Tal-Singer R; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints study investigators. Serum surfactant protein D is steroid sensitive and associated with exacerbations of COPD. Eur Respir J. 2009 Jul;34(1):95-102. doi: 10.1183/09031936.00156508. Epub 2009 Jan 22. PMID 19164344
- [Derived] Lomas DA, Silverman EK, Edwards LD, Miller BE, Coxson HO, Tal-Singer R; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) investigators. Evaluation of serum CC-16 as a biomarker for COPD in the ECLIPSE cohort. Thorax. 2008 Dec;63(12):1058-63. doi: 10.1136/thx.2008.102574. Epub 2008 Aug 29. PMID 18757456
- [Derived] Vestbo J, Anderson W, Coxson HO, Crim C, Dawber F, Edwards L, Hagan G, Knobil K, Lomas DA, MacNee W, Silverman EK, Tal-Singer R; ECLIPSE investigators. Evaluation of COPD Longitudinally to Identify Predictive Surrogate End-points (ECLIPSE). Eur Respir J. 2008 Apr;31(4):869-73. doi: 10.1183/09031936.00111707. Epub 2008 Jan 23. PMID 18216052